CLINICAL TRIAL: NCT05030831
Title: A Phase 1/2, Open-Label, Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of INZ-701 Followed by an Open-Label Long-Term Extension Period in Adults With ABCC6 Deficiency Manifesting as Pseudoxanthoma Elasticum (PXE)
Brief Title: Evaluation of Safety, Tolerability, and Efficacy of INZ-701 in Adults With ABCC6 Deficiency Causing PXE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Inozyme Pharma (Industry)
Collaborators: IQVIA Biotech (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INZ701-201
Record Dates: First submitted 2021-08-26; First posted 2021-09-01 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: ATP-Binding Cassette Subfamily C Member 6 Deficiency; Pseudoxanthoma Elasticum; Generalized Arterial Calcification of Infancy
Keywords: ATP-Binding Cassette Subfamily C Member 6 Deficiency; ABCC6; Pseudoxanthoma elasticum; PXE; Generalized Arterial Calcification of Infancy; GACI; hypopyrophosphatemia
MeSH Terms: conditions — Pseudoxanthoma Elasticum; Arterial calcification of infancy

STUDY DESIGN:
Intervention Model Description: Study INZ701-201 is a Phase 1/2, multicenter, open-label, multiple ascending dose (MAD) study followed by a long-term open-label extension period conducted in adults with ABCC6 Deficiency manifesting as PXE. The study design during the Dose Evaluation Period is a MAD 3+3 with 3 dose cohorts.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- INZ-701 (Experimental): The study design of the Dose Evaluation Period is a MAD 3 + 3 with 3 dose cohorts.
  Based on nonclinical findings and nonclinical pharmacology modeling, the initial planned doses will be 0.2 mg/kg, 0.6 mg/kg, and 1.8 mg/kg, with a twice weekly dose regimen.
  During the Extension Period, INZ-701 administration will initially be at the dose and dose schedule assigned in the Dose Evaluation Period; however, the Sponsor may modify the assigned dose and/or dosing regimen in the Extension Period post-Week 48 based on cumulative review of safety and PK/PD data, including population PK.
  Study visits will be in-clinic every 4 weeks until Week 48 of the Extension Period and then every 12 weeks (remote or in-clinic) until the subject leaves the study. Subjects will complete an End of Study (EOS) Visit (Safety Follow-up Visit) 30 days after their last dose of INZ-701.
  Interventions: Drug: INZ-701

INTERVENTIONS:
Drug: INZ-701 — INZ-701 is a recombinant fusion protein that contains the extracellular domains of human ENPP1 coupled with an Fc fragment from an immunoglobulin gamma-1 (IgG1) antibody (rhENPP1-Fc).
  Other Names: rhENPP1-Fc

SUMMARY:
The purpose of this study is to assess the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics PD) of multiple ascending doses of INZ-701, an ectonucleotide pyrophosphatase/phosphodiesterase 1 (ENPP1) recombinant fusion protein, for the treatment of ABCC6 Deficiency. The goal of the study is to identify a dose regimen for further clinical development in the treatment of ABCC6 Deficiency.

DETAILED DESCRIPTION:
INZ-701 is an ectonucleotide pyrophosphatase/phosphodiesterase 1 (ENPP1) recombinant fusion protein in development for the treatment of ABCC6 Deficiency, a rare genetic disorder.

Study INZ701-201 is a Phase 1/2, multicenter, open-label, multiple ascending dose (MAD), dose-finding study followed by a long-term open-label Extension Period conducted in adults with ABCC6 Deficiency manifesting as Pseudoxanthoma elasticum (PXE). This study is designed to assess the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of multiple ascending doses of INZ-701. The goal of the study is to identify a dose and dose schedule (number of doses per week) for further clinical development in ABCC6 Deficiency. No placebo will be used in this study.

Exploratory endpoints for the Extension Period of the study include evaluations of arterial and organ calcification, ophthalmologic, cardiac and renal parameters, and physical function as well as patient reported outcomes.

Subject participation consists of a Screening Period of up to 60 days, a 32-day Dose Evaluation Period, and an Extension Period during which subjects may continue to receive INZ-701 (with options for self-, caregiver-, or healthcare provider administration) until INZ-701 is approved and available in the country where the subject resides or until an alternative study for subjects to continue receiving study drug is available. During the Extension Period, follow-up visits will be conducted every 4 weeks until Week 48 of the Extension Period and then every 12 weeks (remote or in-clinic) until the subject leaves the study.

Subjects will complete a follow up visit 30 days after their last dose of INZ-701.

ELIGIBILITY:
Inclusion Criteria

Individuals eligible to participate must meet all of the following inclusion criteria:

1. Must provide written or electronic consent after the nature of the study has been explained, and prior to any research-related procedures, per International Conference on Harmonisation (ICH) Good Clinical Practice (GCP)
2. Clinical diagnosis of PXE supported by prior genetic identification of biallelic ABCC6 mutations (ie, homozygous or compound heterozygous)
3. Male or female, 18 to <70 years of age at Screening
4. Plasma PPi <1300 nM at Screening
5. Subjects who are being treated with statins or proprotein convertase subtilisin/kexin type 9 (PCSK9) inhibitors must have been on treatment for at least 6 months prior to Screening and no new anti-lipid therapy can be introduced within 6 months of Screening
6. Women of child-bearing potential (WOCBP) as defined in Clinical Trials Facilitation and Coordination Group (CTFG 2020) must have a negative serum pregnancy test at Screening
7. WOCBP and partners of fertile males who are WOCBP must be using or agree to use one highly effective form of contraception (per CTFG 2020) and a barrier method from at least 1 month before the first dose of INZ-701 through 30 days after the last dose of INZ-701 (greater than 5 half-lives of INZ-701). WOCBP and partners of fertile males who are WOCBP must also agree to not donate ova from the period following the first dose of INZ-701 through 30 days after last dose of INZ-701.
8. Males who are sexually active must agree to use condoms from the period following first dose of INZ-701 through 30 days after the last dose of INZ-701. Males must also agree to not donate sperm from the period following the first dose of INZ-701 through 30 days after last dose of INZ-701.
9. In the opinion of the Investigator, must be willing and able to complete the Dose Evaluation Period
10. Agree to provide access to relevant medical records

Individuals who meet any of the following exclusion criteria will not be eligible to participate:

1. In the opinion of the Investigator, presence of any clinically significant disease (outside of those considered associated with the diagnosis of ABCC6 Deficiency) that precludes study participation or may confound interpretation of study results, including known uncontrolled thyroid, or unrelated connective tissue, bone, mineral, lipid, ophthalmologic, or muscle disease
2. Active retinal bleeding in both eyes during Screening
3. Clinically significant abnormal laboratory result at Screening in the opinion of the Investigator, including but not limited to, estimated glomerular filtration rate (eGFR) <60 mL/min/1.73m2 (Chronic Kidney Disease-Epidemiology Collaboration equation) or 25-hydroxyvitamin D levels <12 ng/mL
4. Known active fungal, bacterial, and/or viral infection including human immunodeficiency virus, hepatitis B virus, hepatitis C virus, or COVID-19 infection.
5. Malignancy within the last 5 years, except non-melanoma skin cancers or cervical carcinoma in situ
6. Known intolerance to INZ-701 or any of its excipients
7. Unable to or unwilling to discontinue the use of any prohibited medication as provided in the protocol. Discontinuation should be undertaken only if considered not detrimental and indicated by the subject's treating physician.
8. Concurrent participation in another non-Inozyme interventional clinical study and/or receipt of any other investigational new drug within 5 half-lives of the last dose of the other investigational drug or from 4 weeks prior to the first dose of INZ-701, whichever is longer, or use of an investigational device through completion of participation in the study
9. Subjects who are pregnant, trying to become pregnant, or breastfeeding
10. Subjects who are trying to father a child

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2024-07-09 (Actual); Study Completion 2024-07-09 (Actual)

PRIMARY OUTCOMES:
Number of Treatment Emergent Adverse Events (TEAEs) | 32 days (Dose Evaluation Period)
  Treatment-emergent AEs are defined as any AE occurring from the first dose of INZ-701 through 30 days after the last dose of INZ-701.
Number of Treatment Emergent Adverse Events (TEAEs) | 52 weeks (Day 1 through Safety Follow-up Visit)
  Treatment-emergent AEs are defined as any AE occurring from the first dose of INZ-701 through 30 days after the last dose of INZ-701.

SECONDARY OUTCOMES:
Incidence of Anti-Drug Antibodies (ADAs) | 32 days (Dose Evaluation Period)
  The presence of ADAs will be assessed and, if present, further evaluation will determine specificity and subtypes.
Incidence of Anti-Drug Antibodies (ADAs) | 52 weeks (Day 1 through Safety Follow-up Visit)
  The presence of ADAs will be assessed and, if present, further evaluation will determine specificity and subtypes.
Area under the Plasma Concentration versus Time Curve (AUC) of INZ-701 | 32 days (Dose Evaluation Period)
  For each subject, variation of concentration of INZ-701 in the plasma will be measured via a series of blood samples obtained throughout the study, comparing the subject's baseline value over time.
Maximum Plasma Concentration (Cmax) of INZ-701 | 32 days (Dose Evaluation Period)
  For each subject, the maximum concentration of INZ-701 in the plasma will be measured via a series of blood samples obtained throughout the study, comparing the subject's baseline value over time.
Systemic Clearance of INZ-701 | 32 days (Dose Evaluation Period)
  For each subject, clearance of INZ-701 from the body will be measured via a series of blood samples obtained throughout the study, comparing the subject's baseline value over time.
Change from Baseline in Plasma Inorganic Pyrophosphate (PPi) Levels | 32 days (Dose Evaluation Period)
  For each subject, plasma PPi will be measured via a series of blood samples obtained throughout the study, comparing the subject's baseline value over time.
Change from Baseline in Plasma Inorganic Pyrophosphate (PPi) Levels | 52 weeks (Baseline through Safety Follow-up Visit)
  For each subject, plasma PPi will be measured via a series of blood samples obtained throughout the study, comparing the subject's baseline value over time.

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Gunter, MD, Study Director — Inozyme Pharma, Inc.
Locations (2):
- Clinilabs, Eatontown, New Jersey, United States
- Richmond Pharmacology Ltd (RPL), London, United Kingdom

IPD SHARING:
Plan to Share IPD: No